CLINICAL TRIAL: NCT02982629
Title: Improving Access to Eye Care in Glaucoma Patients a Prospective, Controlled, Randomized Trial
Brief Title: Improving Access to Eye Care in Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, L. Jay Katz MD, Principal Investigator, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 410005727
Record Dates: First submitted 2015-08-06; First posted 2016-12-05 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Glaucoma
Keywords: Glaucoma; Eye Care; Community Outreach
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Placebo Comparator): Patients in this group do not receive any letters or phone calls after missing follow-up appointment.
  Interventions: Behavioral: Reminder letter Intervention
- Reminder Letter Intervention (Active Comparator): Patients in this group receive letters and phone calls after missing follow-up appointment to reschedule the appointment.
  Interventions: Behavioral: Reminder letter Intervention

INTERVENTIONS:
Behavioral: Reminder letter Intervention — Patients in this group receive letters and phone calls to reschedule missed follow-up appointments.

SUMMARY:
1. To design and develop a prospective, randomized pilot study utilizing information from electronic medical records to address follow-up adherence and reduce the gap between recommended and actual follow-up adherence in patients with glaucoma.
2. To evaluate the impact of a telephone-based intervention on follow-up adherence in patients with glaucoma using a randomly assigned comparison with usual care.

DETAILED DESCRIPTION:
The Wills Eye Health System (WEHS) proposes to conduct a pilot study to evaluate the feasibility and effectiveness of a telephone-based intervention to improve rates of follow-up exams in patients with glaucoma. The prospective, randomized, controlled trial entitled "Improving Access to Eye Care in Patients with Glaucoma" will utilize cohort data from 2013 electronic medical record information to reduce the gap between recommended and actual follow-up utilization of eye care services in glaucoma patients. Patients with glaucoma will be recruited from the Wills Eye Glaucoma clinic who were seen between 3/1/13 and 10/31/13. A recall list will be generated for patients who have scheduled follow-up appointments from 9/1/13 to 11/30/13. These patients will be randomly assigned to the "Usual Care" group or "Intervention" group. The primary outcome will be successful attendance at a follow-up appointment within an appropriate time frame. This intervention is based on a CDC funded project at Wills to improve access to eye care in patients with diabetes. Thus, this pilot study will test the efficacy of a telephone-based intervention to improve follow-up adherence in patients with glaucoma by improving access to eye care.

ELIGIBILITY:
Inclusion Criteria:

* Attended Wills Eye Glaucoma Clinic from 9/1/12 and 10/31/13

Exclusion Criteria:

* Any medical condition that would preclude the subject from providing reliable and valid data.
* Recommended to f/u in less than 1 month time period.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Adherence to Follow-Up | 28 weeks
  Whether patients adhere to follow-up appointments at 28 weeks.

IPD SHARING:
Plan to Share IPD: Yes
A total of 8 papers have been published. Results will be uploaded by 2016.

REFERENCES:
- [Background] Hark LA, Johnson DM, Berardi G, Patel NS, Zeng L, Dai Y, Mayro EL, Waisbourd M, Katz LJ. A randomized, controlled trial to test the effectiveness of a glaucoma patient navigator to improve appointment adherence. Patient Prefer Adherence. 2016 Sep 8;10:1739-48. doi: 10.2147/PPA.S108391. eCollection 2016. PMID 27660423